CLINICAL TRIAL: NCT05449613
Title: Efficacy and Safety Evaluation of Acupoint Application in the Treatment of Knee Osteoarthritis Joint Pain: a Randomized, Double-blind, Controlled Study
Brief Title: Efficacy and Safety Evaluation of Acupoint Application in the Treatment of Knee Osteoarthritis Joint Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Quan Jiang, MD, PhD, Professor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-077-KY
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupoint application (Active Comparator): The acupoint application is applied each stick apply time 2h, once each day. Acupoints selected: Yanglingquan, Dubi, Neixiyan. The treatment lasted for 4 weeks.
  Interventions: Drug: acupoint application
- placebo (Placebo Comparator): The placebo is applied the same acupuncture points, each stick apply time 2h, once each day. Acupoints selected: Yanglingquan, Dubi, Neixiyan. The treatment lasted for 4 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: acupoint application — During the trial, if patients can not tolerate the pain, meloxicam tablets can be added temporarily, and the total amount of medication for each patient during the observation period was recorded.
  Arms: acupoint application
Other: placebo — During the trial, if patients can not tolerate the pain, meloxicam tablets can be added temporarily, and the total amount of medication for each patient during the observation period was recorded.
  Arms: placebo

SUMMARY:
To evaluate the efficacy and safety of acupoint application of Traditional Chinese medicine in the treatment of KOA joint pain through a prospective, randomized, double-blind, placebo-controlled clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Western medicine diagnosed as knee osteoarthritis, clinical classification is primary, and conforms to the TCM syndrome of cold and wet obstruction;
2. Guidelines for the diagnosis and treatment of osteoarthritis 2018 criteria and Kellgren -Lawrence<Ⅲ;
3. VAS pain score ≥40mm (select the limb with the most obvious pain symptom);
4. For patients taking nonsteroidal drugs or other disease-improving drugs (such as cartilage protectants), the dose has been stable for at least 4 weeks;
5. Signed informed consent.

Exclusion Criteria:

1. Patients who underwent intra-articular therapy within 3 months prior to the trial or required relevant surgical treatment within 1 year；
2. Glucocorticoid and joint cavity injection were used 4 weeks before treatment;
3. swelling and heat of knee joint;
4. other diseases causing knee pain; Such as acute joint injury, tuberculous arthritis, rheumatoid arthritis, rheumatoid arthritis, suppurative arthritis, osteomyelitis, psoriatic arthritis, gout, villi nodular synovitis.
5. History or evidence of any of the following diseases during the screening period: serious cardiovascular and cerebrovascular diseases, active or recurrent ulcer of digestive system or other diseases at risk of bleeding, other serious diseases of digestive system, combined with malignant tumor, serious or progressive diseases of blood system or other systems.
6. Patients with other mental diseases who are unable to cooperate or unwilling to cooperate.
7. Before screening, any of the laboratory test indicators met the following criteria: ALT and AST > 1.5 times the upper limit of normal value, Cr > 1.2 times the upper limit of normal value, and other clinically significant laboratory test abnormalities, which were determined by the investigator to be unsuitable for inclusion in the group.
8. allergic constitution or allergic to test drugs, excipients or similar ingredients.
9. Suspected or confirmed history of alcohol or drug abuse;
10. pregnant or lactating women or those who have planned pregnancy recently and do not want to use contraception;
11. Participants in other clinical trials within 3 months prior to enrollment;
12. The investigator considered that the patients should not participate in the clinical trial.Other requirements for inclusion are willingness to participate for the duration of the trial. All patients will receive verbal and written information about the trial and sign a consent form before inclusion. The researcher obtains written consent before inclusion and randomisation.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes in VAS pain score from baseline 4 weeks | 4 weeks
  After treatment.researchers and investigators were assessed by VAS score (0-10cm) for the overall condition of the disease. Participants rated their current state of control from "very good" to "very poor." The researchers rated disease activity status from "no active rheumatism" to "most severe active rheumatism." The score is accurate to one decimal place.

SECONDARY OUTCOMES:
Changes in WOMAC scale scores from baseline | 4 weeks
Health Measurement Scale (SF-36) | 4 weeks
Number of Participants With Metabolic Abnormal Events at All Assessment Time Points. | 4 weeks
  The participants were tested with blood lipid [liver and kidney function [aspartate aminotransferase(AST), alanine aminotransferase(ALT), Urea(Ur), Crea(Cr)] for regular metabolic function evaluation .The number of participants experiencing metabolic abnormal events have been reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China